CLINICAL TRIAL: NCT00198510
Title: Phase III Safety and Efficacy Study of Vitrase (Ovine Hyaluronidase) for Ophthalmic Intravitreal Injection for Clearance of Severe Vitreous Hemorrhage
Brief Title: Safety and Efficacy Study of Vitrase for Clearance of Severe Vitreous Hemorrhage
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VIT-02-08961X
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2013-03-15 (Estimated); Status verified 2013-03

CONDITIONS: Vitreous Hemorrhage; Diabetic Retinopathy
MeSH Terms: conditions — Vitreous Hemorrhage; Diabetic Retinopathy | interventions — Chondroitinases and Chondroitin Lyases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitrase (Experimental): A single dose of 0.05 cc of Vitrase (hyaluronidase) for ophthalmic intravitreal injection is injected into the vitreous chamber.
  Interventions: Drug: Vitrase
- Observation (No Intervention): Observation only, no medication or intravitreal injection

INTERVENTIONS:
Drug: Vitrase — 7.5 IU of Vitrase
  Other Names: ovine hyaluronidase
  Arms: Vitrase
Drug: Vitrase — 55 IU of Vitrase
  Other Names: ovine hyaluronidase
  Arms: Vitrase
Drug: Vitrase — 75 IU of Vitrase
  Other Names: ovine hyaluronidase
  Arms: Vitrase

SUMMARY:
The purpose of this study is to determine if intravitreal injection of Vitrase (ovine hyaluronidase) clears vitreous hemorrhage

ELIGIBILITY:
Inclusion Criteria:

* Severe vitreous hemorrhage that obscures visualization of the fundus on indirect ophthalmoscopy, that has been present >/= 1 month by history or exam
* BCVA is worse than 20/200 at time of screening

Exclusion Criteria:

* Corneal or lenticular abnormalities that preclude fundus observation
* Ongoing ocular infection, inflammation or history of herpetic corneal lesion
* Current or prior retinal detachment or retinal tears or breaks or intraocular tumor
* More than 1 severe vitreous hemorrhage within 6 months
* Previous vitrectomy for any reason
* Hemorrhage is exclusively pre-retinal, or old & organized
* Prior Vitrase for intravitreal injection in either eye
* No light perception in either eye at any time
* Known contraindications to study medication
* Sickle cell disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750
Dates: Start 1998-11; Primary Completion 2001-09 (Actual); Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
Resolution of Vitreous Hemorrhage | 3 months
  Laser treatment of underlying cause of vitreous hemorrhage, or other surgical treatment, or documented evidence of macula & at least 180 degrees of vitreous base, that vitreous hemorrhage cause is resolved

SECONDARY OUTCOMES:
Incidence of complications & adverse events | 12 months
Visual Acuity | 3 months, 6 months, 12 months
  Best correct visual acuity (BCVA)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa R Grillone, PhD, Study Director — ISTA Pharmaceuticals, Inc.
Locations (73):
- United States (61):
  - Retina Centers, PC, Tucson, Arizona
  - Retina Vitreous Associates Medical Group, Beverly Hills, California
  - Maria E. Castillejos, MD, Chula Vista, California
  - Natural Vision, Fresno, California
  - Eye Medical Center of Fresno, Fresno, California
  - Jerry Sebag, MD, Huntington Beach, California
  - University of California, Irvine, Irvine, California
  - California VitreRetinal Center, Menlo Park, California
  - Southern California Desert Retina Consultants, Palm Springs, California
  - Retinal Consultants, Sacramento, California
  - H. Richard McDonald, MD, San Francisco, California
  - Santa Clara Valley Medical Centre, San Jose, California
  - Robert L. Avery, MD, Santa Barbara, California
  - Olive View/UCLA Medical Center, Sylmar, California
  - Retina Consultants of Southern Colorado, Colorado Springs, Colorado
  - University of Colorado Health Sciences Center, Denver, Colorado
  - Danbury Eye Physicians & Surgeons, Danbury, Connecticut
  - New England Retina Associates, Hamden, Connecticut
  - Florida Eye Clinic, Altamonte Springs, Florida
  - Eye Centers of Florida, Fort Myers, Florida
  - Sarasota Retina Institute, Sarasota, Florida
  - Scott E. Pautler, MD, Tampa, Florida
  - Retina Center at Pali Momi, ‘Aiea, Hawaii
  - Illinois Retina Associates SC, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - American Eye Institute, New Albany, Indiana
  - Felix N. Sabates Eye Associates, Prairie Village, Kansas
  - King Y. Lee, MD, Shawnee Mission, Kansas
  - Kurt A. Gitter, MD, New Orleans, Louisiana
  - Retina Specialists, Baltimore, Maryland
  - Wilmer Eye Institute/Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Retina Consultants, PC, Bethesda, Maryland
  - Schepens Retina Associates, Boston, Massachusetts
  - VitreoRetinal Associates, Grand Rapids, Michigan
  - Retina Center PA, Minneapolis, Minnesota
  - Hunkeler Eye Centers, Kansas City, Missouri
  - Retina Associates of Kansas City, Kansas City, Missouri
  - The Center for Advanced Medicine/Barnes Retina Institute, St Louis, Missouri
  - Robert Wood Johnson Medical School/Retina Vitreous Center, New Brunswick, New Jersey
  - Retina Associates of New Jersey, Teaneck, New Jersey
  - Long Island Vitreo Retinal Consultants, Great Neck, New York
  - Ronni M. Lieberman, MD, New York, New York
  - Retina Vitreous Surgeons of Central NY, Syracuse, New York
  - Charlotte Eye, Ear, Nose & Throat Association, Charlotte, North Carolina
  - Carolina Eye Associates, PA, Raleigh, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Retina Associates of Cleveland, Cleveland, Ohio
  - Retina Consultants, Ohio State University, Columbus, Ohio
  - Dean A. McGee Eye Institute, Oklahoma City, Oklahoma
  - Scheie Eye Institute, Philadelphia, Pennsylvania
  - Retina Research of Wills Eye Hospital, Philadelphia, Pennsylvania
  - Carim Eye & Retina Center, Wyomissing, Pennsylvania
  - Southeastern Retina Associates, PC, Knoxville, Tennessee
  - Retina-Vitreous Associates, Nashville, Tennessee
  - Retinal Vascular Center, Houston, Texas
  - Cullen Eye Institute/Baylor College of Medicine, Houston, Texas
  - Valley Retina Institute, PA, McAllen, Texas
  - John Moran Eye Center, Salt Lake City, Utah
  - Vista Retinal Consultants, Roanoke, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (9):
  - Vancouver Eye Care Center/University of British Columbia, Vancouver, British Columbia
  - Dalhousie University, Halifax, Nova Scotia
  - Ivey Institute of Ophthalmology, London, Ontario
  - University of Ottawa Eye Institute, Ottawa, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - Royal Victoria Hospital, Montreal, Quebec
  - Centre Hospitalier de l'Universite Laval (CHUL), Sainte-Foy, Quebec
  - The Medical Centre Pasqua Hospital, Regina, Saskatchewan
  - Saskatoon City Hospital, Saskatoon, Saskatchewan
- Mexico (3):
  - Instituto de Oftalmologia, Fundacion Conde de Valenciana, Col. Obrera, Mexico City
  - Association Para Evitar la Ceguera en Mexico, Coyacan, Mexico City
  - Fundacion Hospital, Nuestra Senora de la Luz IAP, Cuahtemoc, Mexico City

REFERENCES:
- [Derived] Bhavsar AR, Grillone LR, McNamara TR, Gow JA, Hochberg AM, Pearson RK; Vitrase for Vitreous Hemorrhage Study Groups. Predicting response of vitreous hemorrhage after intravitreous injection of highly purified ovine hyaluronidase (Vitrase) in patients with diabetes. Invest Ophthalmol Vis Sci. 2008 Oct;49(10):4219-25. doi: 10.1167/iovs.07-1602. Epub 2008 Apr 25. PMID 18441312